CLINICAL TRIAL: NCT01200264
Title: Open-Label Study to Assess the Safety and Efficacy of Apremilast in Patients With Chronic Plaque Psoriasis Who Have Failed One Course of Biologic Therapy.
Brief Title: Apremilast for Chronic Plaque Psoriasis (CPP) Patients Who Have Failed One Course of Biologic Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Contract never executed; withdrawn by sponsor
Sponsor: Duke University (Other)
Responsible Party: John C. Murray, MD, Professor of Medicine, Duke University Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00025452; AP00039
Record Dates: First submitted 2010-09-10; First posted 2010-09-13 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2010-09

CONDITIONS: Chronic Plaque Psoriasis
MeSH Terms: interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- apremilast for all subjects (Experimental)
  Interventions: Drug: apremilast

INTERVENTIONS:
Drug: apremilast — apremilast 10 mg tablets with dose titration to 30 mg BID for 169 days
  Other Names: CC-1004

SUMMARY:
This is a Phase II, open label, investigator-initiated study to be done at Duke University Medical Center to treat adult patients (ages 18-80) with chronic plaque psoriasis who have failed Biologic Therapy with Apremilast 30 mg BID for 24 weeks. At the time of enrollment, the patient must have received biologic therapy without achieving a response of "almost clear" or "clear" according to PGA or has not responded with a 75% reduction of PASI score. Once deemed eligible, subjects will return for a baseline visit and receive Apremilast therapy and instructions. Subjects will be treated at weeks 0,4,8,12,16,20 and 24; subjects will be evaluated 28 days after last dose of Apremilast for safety and efficacy.

DETAILED DESCRIPTION:
Data Analysis Data will be analyzed and reported after all subjects have completed follow-up phase of study. All subsequent data collected will be analyzed and reported in a follow-up clinical report.

Data & Safety Monitoring Dr. Murray will be following all laboratory values and adverse events during this trial. In addition, Celgene will provide a study monitor to, at regular intervals, review all data. All data will be reported to Celgene.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18-80 yrs diagnosed with moderate-to-severe chronic plaque psoriasis with a PGA of 3 or greater and require systemic therapy
* Must have received a biologic therapy for CPP and did not achieve a PGA of 'almost clear' or 'clear'
* Must meet lab criteria per Pg 20-21 of protocol
* All subjects must follow contraceptive measures as described in protocol, Pg 21.

Exclusion Criteria:

* Abnormal Chest x-ray
* Significant abnormality of ECG
* Positive HIV Ab, Hepatitis B & C
* Subjects with erythrodermic, pustular or guttate psoriasis are ineligible
* Serious local infection or systemic infection, or tuberculosis within 3 mos of first dose of apremilast

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2011-12 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Safety/efficacy of apremilast in CPP pts that have failed 1 course of biologic therapy | 6 mos. treatment and 1 month F/U post treatment

SECONDARY OUTCOMES:
Mechanistic studies performed to assess efficacy of apremilast to inhibit inflammatory responses in non-involved, mildly traumatized skin. | Treatment course of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: John C Murray, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States